CLINICAL TRIAL: NCT01214018
Title: Evaluation of Post-traumatic Stress Among the Nearest Relatives of Brain-dead Organ Donors: Comparison With the Nearest-relatives of Brain-dead Patients Who Were Not Organ Donors for Medical or Legal Reasons, or Because of Donation Opposition
Brief Title: Evaluation of Post-traumatic Stress Among the Nearest Relatives of Brain-dead Organ Donors
Status: Terminated | Type: Observational
Why Stopped: No recruitment
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2009/CB-04
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Stress Disorders, Post-Traumatic; Tissue Donors; Tissue and Organ Procurement
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Reference: Nearest relatives of brain-dead patients who donated organs
  Interventions: Other: Questionnaires and interview
- Opposition: Nearest relatives of brain-dead patients opposed to organ donation
  Interventions: Other: Questionnaires and interview
- Medical/Legal: Nearest relatives of brain-dead patients for whom organ donation was not an option because of medical or legal reasons
  Interventions: Other: Questionnaires and interview

INTERVENTIONS:
Other: Questionnaires and interview — Questionnaires and interview

SUMMARY:
The goal is to compare post tramautic stress between the nearest relatives of brain-dead patients who are organ donor to those of brain-dead patients who are not organ donors for medical, legal or opposition reasons.

ELIGIBILITY:
Inclusion Criteria:

* must be one of the following: person-of-trust previously designated by the deceased, a spouse, sibling, parent, or child of the deceased

Exclusion Criteria:

* refusal to participate
* does not speak French
* deaf/mute
* adult, but under guardianship

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants are the nearest relatives of brain-dead patients
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2011-05-15 (Actual); Primary Completion 2016-05-15 (Actual); Study Completion 2016-05-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with an IES score > 37 | 2 hours
  The IES score follows Azoulay et al (2005). Am J Respir Crit Care Med. 171: 987-94. IES = Impact of Event Scale - revised, ranging from 0 to 88, with 88 being the greatest risk for post-traumatic stress

SECONDARY OUTCOMES:
The IES score | 2 hours
  The Impact of Event Scale - revised, ranging from 0 to 88
Hospital Depression and Anxiety Score (HDAS) | 2 hours
  score ranging from 0 (no symptoms) to 21 (max). HDAS scores >=8 indicate clinically significant depression or axiety

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Boutin, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (4):
- France (4):
  - CH Henry Duffaut, Avignon
  - Centre Hospitalier Général, Béziers
  - Hôpital Guy de Chauliac, CHU de Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nîmes, Nîmes